CLINICAL TRIAL: NCT00048412
Title: Phase I/II Study of Allogeneic Stem Cell Transplantation for Patients With Hematologic Malignancy, Using MHC Identical or Near Identical Donors and Sub-Myeloablative Conditioning With CAMPATH 1H (DIMSUM)
Brief Title: Stem Cell Transplant for Patients With Blood Malignancy Using Donors and Less Toxic Chemotherapy With CAMPATH 1H
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: The Methodist Hospital Research Institute (Other); Center for Cell and Gene Therapy, Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, George Carrum, Professor, Baylor College of Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H8714; DIMSUM
Record Dates: First submitted 2002-10-30; First posted 2002-11-01 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Myelodysplastic Disorders; Leukemia; Multiple Myeloma; Plasma Cell Dyscrasia; Lymphoproliferative Disorders
MeSH Terms: conditions — Leukemia; Multiple Myeloma; Paraproteinemias; Lymphoproliferative Disorders | interventions — fludarabine; Alemtuzumab

INTERVENTIONS:
Drug: FLUDARABINE
Drug: CAMPATH 1H
Drug: FK50
Procedure: Stem Cell Collection and Infusion

SUMMARY:
1. To assess the treatment related mortality of allogeneic stem cell transplantation with non-myeloablative therapy incorporating the lymphodepleting MAb CAMPATH-1H, in patients with hematological diseases and renal cell carcinoma not eligible for conventional (myeloablative) therapy.
2. To assess the time to engraftment and incidence of graft failure in patients receiving this transplant regimen.
3. To assess the safety, pharmacokinetics and immunologic activity of CAMPATH-1H when used as part of a subablative conditioning regimen.

DETAILED DESCRIPTION:
This is a two arm study in which outcomes will be assessed independently in recipients of HLA matched sibling transplants and recipients of unrelated or mismatched family donor transplants, although both groups will receive identical treatments.

The following will be given to the patient after admission:

Day - 6: Total body irradiation

Day - 5 to - 2: Fludarabine and Campath 1H

Day - 1: Day of rest

Day 0: Stem cell transplant (infusion)

ELIGIBILITY:
Inclusion criteria

1. Diagnosis of myelodysplastic disorders, Acute Myelogenous Leukemia, Acute Lymphoblastic Leukemia, Multiple Myeloma, Plasma Cell Dyscrasia, Lymphoproliferative disorders (Non-Hodgkin Lymphoma, Hairy Cell Leukemia, Chronic Lymphocytic Leukemia and Hodgkins Disease) or Renal Cell Carcinoma.
2. Conditions that increase treatment related mortality (need one or more to be eligible):

   1. Greater to or equal to 50 years of age.
   2. EF of less than 45%
   3. DLCO less than 50% of FEV1 50-75% of predicted value.
   4. Diabetes Mellitus
   5. Renal Insufficiency (but creatine clearance not less than 25ml/min).
   6. Prior recent history of systemic fungal infection.
   7. 3rd or greater remission of AML or ALL
   8. More than 1 year of diagnosis (CML or Myeloma patients)
   9. Multiple types of treatment regimens. (equal to or more than 3)
   10. Prior autologous or allogeneic stem cell transplantation.
   11. Significant grade III or IV neurologic or hepatic toxicity from previous treatment.
   12. No matched sibling donor.
3. Available healthy donor without any contraindications for donation. 5/6 or 6/6 related donor. 5/6 or 6/6 unrelated donor (molecular typing for DRB1)
4. Patient and/or responsible person able to understand consent.
5. Age between birth and 70 years.
6. For women of childbearing potential, negative pregnancy test.

Exclusion criteria

1. Patient is pregnant, lactating or unwilling to use contraceptives
2. HIV positive patient
3. Uncontrolled intercurrent infection
4. Refractory AML, or ALL
5. Untreated Blast Crisis for CML
6. Uncontrolled High-grade lymphoproliferative disease/lymphoma.
7. Unstable angina and uncompensated congestive heart failure (Zubrod of 3 or greater)
8. Severe chronic pulmonary disease requiring oxygen (Zubrod of 3 or greater)
9. Hemodialysis dependent
10. Active Hepatitis or cirrhosis with total bilirubin, SGOT, and SGPT greater than 3 x normal.
11. Unstable Cerebral vascular disease and recent hemorrhagic stroke (less than 6 months)
12. Active CNS disease from hematological disorder.

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40
Dates: Start 2000-06; Primary Completion 2004-11-12 (Actual); Study Completion 2004-11-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George Carrum, MD, Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - Texas Children's Hospital, Houston, Texas
  - The Methodist Hospital, Houston, Texas